CLINICAL TRIAL: NCT03379675
Title: A Pilot Phase 2a, Randomized, Double-blind, Placebo-controlled Study to Explore the Antiviral Activity, Clinical Outcomes, Safety, Tolerability, and Pharmacokinetics of JNJ-53718678 at Two Dose Levels in Non-Hospitalized Adult Subjects Infected With Respiratory Syncytial Virus
Brief Title: A Study to Explore the Antiviral Activity, Clinical Outcomes, Safety, Tolerability, and Pharmacokinetics of JNJ-53718678 at Two Dose Levels in Non-Hospitalized Adult Participants Infected With Respiratory Syncytial Virus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108419; 2017-003252-24 (EudraCT Number); 53718678RSV2004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-12-15; First posted 2017-12-20 (Actual); Results first posted 2022-06-28 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — JNJ-53718678

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A: JNJ-53718678 500 mg (Experimental): Participants will receive 500 mg dose of JNJ-53718678 once daily for 7 days.
  Interventions: Drug: JNJ-53718678 500 mg
- Treatment B: JNJ-53718678 80 mg + Placebo (Experimental): Participants will receive 80 mg dose of JNJ-53718678 along with the matching placebo to the same total volume as for the 500 mg dose once daily for 7 days.
  Interventions: Drug: JNJ-53718678 80 mg; Drug: Placebo
- Treatment C: Placebo (Placebo Comparator): Participants will receive matching placebo to the same total volume as for the 500 mg dose once daily for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-53718678 500 mg — Participants will receive 500 mg dose of JNJ-53718678 oral solution once daily for 7 days.
  Arms: Treatment A: JNJ-53718678 500 mg
Drug: JNJ-53718678 80 mg — Participants will receive 80 mg dose of JNJ-53718678 oral solution along with the matching placebo to the same total volume as for the 500 mg dose once daily for 7 days.
  Arms: Treatment B: JNJ-53718678 80 mg + Placebo
Drug: Placebo — In treatment B, participants will receive matching placebo along with JNJ-53718678 to maintain the same total volume as for the 500 mg dose once daily for 7 days. In treatment C, participants will receive matching placebo to the same total volume as for the 500 mg dose once daily for 7 days.
  Arms: Treatment B: JNJ-53718678 80 mg + Placebo; Treatment C: Placebo

SUMMARY:
The purpose of this study is to explore the antiviral effect of JNJ-53718678 at 2 dose levels (80 milligrams [mg] and 500 mg) once daily for 7 days in adults with Respiratory Syncytial Virus (RSV) infection, as measured by RSV viral load in nasal secretions by quantitative reverse transcription polymerase chain reaction (qRT-PCR) assay.

DETAILED DESCRIPTION:
This study will be performed to explore the antiviral activity, clinical outcomes, safety, tolerability, and pharmacokinetics of JNJ-53718678 in adult participants infected with RSV. The study will include both participants who are otherwise healthy (ie, without underlying condition) or who have comorbid conditions (eg, asthma, chronic obstructive pulmonary disease (COPD), cardiovascular disease, other chronic diseases), with the exception of immunocompromised participants, presenting for medical care but not requiring hospitalization. The study will include a screening period (Day -1 to Day 1), a treatment Period (Day 1 to Day 8), and a follow-up period (Day 9 to Day 28). Safety evaluations will include adverse events, laboratory tests, electrocardiogram, vital signs, physical examination, and specific toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have an acute respiratory illness with signs and symptoms consistent with a viral infection (example, fever, cough, nasal congestion, runny nose, sore throat, myalgia, lethargy, shortness of breath, or wheezing) with onset less than or equal to 5 days from the anticipated time of randomization. Onset of symptoms is defined as the time the participant becomes aware of the first sign and/or symptom consistent with a viral infection
* Participant has been diagnosed with respiratory syncytial virus (RSV) infection using a rapid polymerase chain reaction (PCR) based or rapid-antigen-detection test
* Before randomization, a woman must be not of childbearing potential defined as: Premenarchal, Postmenopausal or Permanently sterile
* A male participant must agree to the use of acceptable contraceptive measures
* With the exception of the RSV-related illness the participant must be medically stable on the basis of physical examination, medical history, vital signs, and electrocardiogram (ECG) performed at screening

Exclusion Criteria:

* Hospitalized participants or participants expected to be hospitalized within 24 hours of screening
* History of or concurrent illness (beyond a comorbid condition) that in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant or that could prevent, limit, or confound the protocol-specified assessments
* Participants who had major surgery within the 28 days prior to randomization or have planned major surgery through the course of the study
* Participants who are considered by the investigator to be immunocompromised within the past 12 months
* Participant has known or suspected chronic or acute hepatitis B or C infection
* Women who are pregnant or breastfeeding
* Participants with clinically significant abnormal ECG findings (other than QT-interval corrected for heart rate according to Fridericia [QTcF] interval greater than [>] 500 millisecond [ms]) not consistent with the underlying condition in the study population, as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (124):
- United States (13):
  - Core Healthcare Group, Cerritos, California
  - eStudySite, Chula Vista, California
  - SC Clinical Research Inc, Garden Grove, California
  - Lake Internal Medicine Associates, Eustis, Florida
  - Florida Research Center Inc., Miami, Florida
  - Family Medicine, Nampa, Idaho
  - William Beaumont Hospital, Royal Oak, Michigan
  - AllinaHealth - Abbott Northwestern Hospital (13520), Minneapolis, Minnesota
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - Onsite Clinical Solutions, Charlotte, North Carolina
  - Unity Clinical Research, Lindsay, Oklahoma
  - Spectrum Medical Research, Gaffney, South Carolina
  - Fusion Clinical Research of Spartanburg, Spartanburg, South Carolina
- Argentina (12):
  - Hospital Espanol De Bahia Blanca, Bahía Blanca
  - Hospital Interzonal General de Agudos Dr. Jose Penna, Bahía Blanca
  - Hospital Privado - Centro Medico de Cordoba, Barrio Parque Velez Sarfield
  - Fundación Respirar, CABA
  - Hospital Italiano de La Plata, Ciudad de La Plata
  - HIGA Prof. Dr. Ramón Carrillo, Ciudadela
  - Hospital Rawson, Córdoba
  - Hospital Italiano de Cordoba, Córdoba
  - Hospital Cordoba, Córdoba
  - Sanatorio Juan XXIII, General Roca
  - Instituto Médico de la Fundación de Estudios Clínicos (ECLIN), Rosario
  - Clinica Mayo de UMCB, San Miguel de Tucumán
- Australia (6):
  - Paratus Clinical Blacktown Clinic, Blacktown
  - Barwon Health - University Hospital Geelong, Geelong
  - Paratus Clinical Kanwal Clinic, Kanwal
  - Paratus Clinical Kippa Ring Clinic, Kippa-Ring
  - Mater Hospital Brisbane, South Brisbane
  - Westmead Hospital, Sydney
- Belgium (4):
  - CHU Saint-Pierre, Brussels
  - Jaak Mortelmans, Ham
  - BVBA Dr. Luc Capiau, Massemen
  - Testumed, Tessenderlo
- Brazil (10):
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte
  - Fundacao para o Desenvolvimento Medico Hospitalar (UNESP Botucatu), Botucatu
  - Universidade Federal de Santa Catarina, Florianópolis
  - Centro de Estudos e Pesquisas em Moléstias Infecciosas - CEPCLIN, Natal
  - Associacao Hospitalar Beneficente Sao Vicente de Paulo - Hospital Sao Vicente de Paulo, Passo Fundo
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da PUCRS, Porto Alegre
  - Universidade Federal da Bahia - Hospital Professor Edgard Santos, Salvador
  - Sociedade Beneficente de Senhoras - Hospital Sírio Libanês, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - Hospital Heliopolis, São Paulo
- Bulgaria (6):
  - MHAT 'Sv. Ivan Rilski' Kozloduy EOOD, Kozloduy
  - Specialized Hospital for Active Treatment of Pulmonary Diseases - Pernik, Pernik
  - SHAT of Pneumo-phthisiatric Diseases Dr Dimitar Gramatikov - Ruse, EOOD, Rousse
  - MHAT 'Dr. Bratan Shukerov', Smolyan
  - Diagnostic Consultation Centre 'Alexandrovska' EOOD, Sofia
  - Specialized Hospital for Active Treatment of Pulmonary Diseases - Troyan EOOD, Troyan Municipality
- Canada (4):
  - Aggarwal and associates Ltd, Brampton, Ontario
  - Milestone Research, London, Ontario
  - Dr Anil K Gupta Medicine Professional Corporation, Toronto, Ontario
  - Clinique Force Medic (GCP Trials), Montreal, Quebec
- France (6):
  - Centre Hospitalier d'Agen, Agen
  - Cabinet du Dr Remaud, Angers
  - Maison Medicale Rive Sud, Mûrs-Erigné
  - CHU Nantes - Hotel Dieu, Nantes
  - Cabinet du Dr Boye, Nantes
  - Cabinet du Dr Baranes, Paris
- Germany (4):
  - MECS GmbH, Berlin
  - IKF Pneumologie GmbH & Co. KG Am Standort IFS - Interdisziplinäres Facharztzentrum, Frankfurt
  - Klinische Forschung Hannover-Mitte GmbH, Hanover
  - Hausarztpraxis am Lindenplatz, Lübeck
- Japan (10):
  - Fukui General Clinic, Fukui-shi
  - Koukan Clinic, Kawasaki
  - Shinkomonji hospital, Kitakyushu
  - Musashikoganei Clinic, Koganeishi
  - Medical Square Kuhonji Clinic, Kumamoto
  - Rinku General Medical Center, Osaka
  - Tokyo Shinagawa Hospital, Shinagawa-ku
  - Saino Clinic, Tokorozawa-shi
  - Toyota Kosei Hospital, Toyota
  - Shin Yukuhashi Hospital, Yukuhashi
- Mexico (5):
  - Hospital Cardiologica Aguascalientes, Aguascalientes
  - Centro de Investigacion Medico Biologica y Terapia Avanzada CIMBYTA, Guadalajara
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara
  - RM Pharma Specialists, México
  - Hospital Universitario de Nuevo Leon 'Dr Jose Eleuterio Gonzalez', Monterrey
- Poland (6):
  - Indywidualna Specjalistyczna Praktyka Lekarska Lek. Krzysztof Lis, Kielce
  - Centrum Medyczne All Med, Krakow
  - Diamond Clinic, Krakow
  - SPZOZ Uniwersytecki Szpital Kliniczny nr 1 im.Barlickiego Uniwersytetu Med. w Lodzi Zespol Poradni, Lodz
  - Beata Asankowicz-Bargiel i Partnerzy, Lekarze-sp. Spec. Poradnia Pulmonologiczna, Ostrów Wielkopolski
  - Centrum Badan Klinicznych, Osrodek Badan Wczesnej Fazy, Wroclaw
- Russia (5):
  - Krasnogorsk city hospital #1, Krasnogorsk
  - City Polyclinic #25 of the Nevsky District of SPB, Saint Petersburg
  - LLC 'Medical centr 'Reavita Med Spb', Saint Petersburg
  - Eco-safety Ltd, Saint Petersburg
  - Research Institute of Influenza, Saint Petersburg
- South Africa (4):
  - Soweto Clinical Trial Centre, Johannesburg
  - Newtown Clinical Research, Johannesburg
  - Emmed Research, Pretoria
  - Welkom Clinical Trial Centre, Welkom
- South Korea (7):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Kyungpook National University Hospital, Daegu
  - The Catholic university of Korea, St. Vincent's Hospital, Gyeonggi-do
  - Gachon University Gil Hospital, Incheon
  - Inha University Hospital, Incheon
  - Kangnam Sacred Heart Hospital, Seoul
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul
- Spain (6):
  - Hosp. Gral. Univ. de Alicante, Alicante
  - Hosp. Gral. Univ. de Elche, Elche
  - Hosp. Univ. Virgen de Las Nieves, Granada
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
  - Hosp. Alvaro Cunqueiro, Vigo
- Sweden (3):
  - Skanes universitetssjukhus, Malmo
  - Norrlands Universitetssjukhus, Umeå
  - Akademiska Sjukhuset, Uppsala
- Taiwan (5):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - Kuang Tien General Hospital- Dajia, Taichung
  - Taipei Municipal Wanfang Hospital, Taipei
  - Far Eastern Memorial Hospital, Taipei
- Ukraine (8):
  - Medical Center of LL Company 'Scientific Medical Center-Your Doctor', Kharkiv
  - Medical Unit Of Company 'Kharkiv Tractor Plant', Kharkiv Medical Academy Of Postgraduate Education, Kharkiv
  - Mi 'Kherson City Clinical Hospital Of E.E. Karabelesh', Kherson
  - Kyiv Railway Clinical Hospital #2 Of Branch 'Health Center' Of The Company 'Ukrainian Railway', Kyiv
  - Policlinic of State Joint Stock Holding Company 'Artem', Kyiv
  - Private Small Enterprise Medical Center Pulse, Vinnytsia
  - Medical Center Ltd 'Health Clinic', Department Of General Therapy, Vinnytsia
  - Vinnytsia City Clinical Hospital #1, Vinnytsia National Medical University, Vinnytsia

REFERENCES:
- [Derived] Nilsson AC, Pullman J, Napora P, Luz K, Gupta A, Draghi J, Guzman Romero AK, Aggarwal N, Petrova G, Ianus J, Vijgen L, Scott J, Sinha R, Rusch S, Huntjens D, Bertzos K, Stevens M; ROSE Study Group. A pilot phase 2a, randomized, double-blind, placebo-controlled study to explore the antiviral activity, clinical outcomes, safety, and tolerability of rilematovir at two dose levels in non-hospitalized adults with respiratory syncytial virus infection. Clin Microbiol Infect. 2023 Oct;29(10):1320-1327. doi: 10.1016/j.cmi.2023.07.004. Epub 2023 Jul 6. PMID 37422079

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment A: JNJ-53718678 500 mg: Participants received JNJ-53718678 500 milligrams (mg) as an oral solution once daily for 7 days.
- Treatment B: JNJ-53718678 80 mg + Placebo: Participants received JNJ-53718678 80 mg as an oral solution once daily for 7 days. In addition, participants received matching placebo to maintain the blinding.
- Treatment C: Placebo: Participants received matching placebo as an oral solution once daily for 7 days.
Period: Overall Study
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Started | 24 | 24 | 24
Completed | 20 | 22 | 22
Not Completed | 4 | 2 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo | Total
Number analyzed (Participants) | 24 | 24 | 24 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (17.89) | 48.4 (17.39) | 58.9 (14.16) | 53 (16.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 14 | 37
  Male | 12 | 13 | 10 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 8 | 23
  Not Hispanic or Latino | 17 | 16 | 15 | 48
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 1 | 2 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 3
  White | 21 | 20 | 19 | 60
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 4 | 3 | 5 | 12
  Belgium | 0 | 0 | 1 | 1
  Brazil | 1 | 3 | 1 | 5
  Bulgaria | 2 | 3 | 2 | 7
  Canada | 4 | 3 | 3 | 10
  France | 0 | 0 | 1 | 1
  Germany | 3 | 0 | 3 | 6
  Mexico | 2 | 2 | 2 | 6
  Poland | 3 | 3 | 2 | 8
  Russia | 0 | 1 | 0 | 1
  Spain | 1 | 0 | 1 | 2
  Taiwan, Province Of China | 0 | 1 | 1 | 2
  Ukraine | 2 | 1 | 0 | 3
  United States | 2 | 2 | 2 | 6
  Sweden | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Respiratory Syncytial Virus (RSV) Viral Load (VL)-Time Curve (AUC) From Immediately Prior to First Dose of Study Drug (Baseline) Through Day 3
Description: Area under the RSV VL-time curve (AUC) was determined as log10 copies*hour per milliliter (Log10 copies*hr/mL) by quantitative reverse transcription polymerase chain reaction (qRT-PCR) assay of mid turbine nasal swabs.
Time Frame: Baseline through Day 3
Population: The intent-to-treat-infected (ITT-i) population consisted of all randomized participants who received at least 1 dose of study drug and who had a central lab-confirmed RSV infection. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Log10 copies*hr/mL
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 21 | 21 | 21
Log10 copies*hr/mL | 207.3 (89.55) | 246.3 (67.39) | 203.4 (87.63)

2. Primary Outcome: Area Under the RSV VL-time Curve (AUC) From Immediately Prior to First Dose of Study Drug (Baseline) Through Day 5
Description: Area under the RSV VL-time curve (AUC) was determined as Log10 copies*hr/mL by qRT-PCR assay of mid turbine nasal swabs.
Time Frame: Baseline through Day 5
Population: The ITT-i population consisted of all randomized participants who received at least 1 dose of study drug and who had a central lab-confirmed RSV infection. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Log10 copies*hr/mL
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 20 | 21 | 21
Log10 copies*hr/mL | 344.5 (189.40) | 424.2 (145.73) | 340.4 (148.30)

3. Primary Outcome: Area Under the RSV VL-time Curve (AUC) From Immediately Prior to First Dose of Study Drug (Baseline) Through Day 8
Description: Area under the RSV VL-time curve (AUC) was determined as Log10 copies*hr/mL by qRT-PCR assay of mid turbine nasal swabs.
Time Frame: Baseline through Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 copies*hr/mL
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 20 | 21 | 21
Log10 copies*hr/mL | 470.7 (305.38) | 612.3 (253.29) | 486.1 (254.15)

4. Primary Outcome: Area Under the RSV VL-time Curve (AUC) From Immediately Prior to First Dose of Study Drug (Baseline) Through Day 14
Description: Area under the RSV VL-time curve (AUC) was determined as Log10 copies*hr/mL by qRT-PCR assay of mid turbine nasal swabs.
Time Frame: Baseline through Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 copies*hr/mL
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 20 | 19 | 20
Log10 copies*hr/mL | 534.4 (379.92) | 747.1 (352.25) | 619.9 (394.15)

5. Primary Outcome: Change From Baseline in RSV Viral Load at Day 3
Description: Change from baseline in RSV viral load at Day 3 was measured as Log10 copies/mL by qRT-PCR assay in the mid-turbinate nasal swab specimens.
Time Frame: Baseline to Day 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 21 | 20 | 20
Log10 copies/mL | -2.210 (1.7185) | -1.436 (1.6165) | -2.221 (1.7093)

6. Primary Outcome: Change From Baseline in RSV Viral Load at Day 5
Description: Change from baseline in RSV viral load at Day 5 was measured as Log10 copies/mL by qRT-PCR assay in the mid-turbinate nasal swab specimens.
Time Frame: Baseline to Day 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 20 | 21 | 21
Log10 copies/mL | -3.156 (2.2887) | -2.324 (1.6727) | -3.031 (1.5010)

7. Primary Outcome: Change From Baseline in RSV Viral Load at Day 8
Description: Change from baseline in RSV viral load at Day 8 was measured as Log10 copies/mL by qRT-PCR assay in the mid-turbinate nasal swab specimens.
Time Frame: Baseline to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 22 | 21 | 21
Log10 copies/mL | -4.960 (1.7804) | -3.983 (1.3928) | -3.953 (1.5674)

8. Primary Outcome: Change From Baseline in RSV Viral Load at Day 14
Description: Change from baseline in RSV viral load at Day 14 was measured as Log10 copies/mL by qRT-PCR assay in the mid-turbinate nasal swab specimens.
Time Frame: Baseline to Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 22 | 21 | 21
Log10 copies/mL | -5.135 (1.6444) | -5.777 (1.6183) | -4.858 (1.7419)

9. Primary Outcome: Change From Baseline in RSV Viral Load at Day 21
Description: Change from baseline in RSV viral load oat Day 21 was measured as Log10 copies/mL by qRT-PCR assay in the mid-turbinate nasal swab specimens.
Time Frame: Baseline to Day 21
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 22 | 21 | 21
Log10 copies/mL | -5.433 (2.1416) | -5.898 (1.6421) | -5.129 (1.6513)

10. Primary Outcome: RSV Viral Load at Baseline
Description: RSV viral load was measured as log10 copies/mL by qRT-PCR assay in the mid-turbinate nasal swab specimens.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 23 | 21 | 22
Log10 copies/mL | 5.523 (1.7911) | 5.851 (1.6777) | 5.285 (1.7158)

11. Primary Outcome: RSV Viral Load at Day 3
Description: RSV viral load was measured as log10 copies/mL by qRT-PCR assay in the mid-turbinate nasal swab specimens.
Time Frame: Day 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 21 | 20 | 20
Log10 copies/mL | 3.267 (2.5490) | 4.448 (1.9513) | 3.160 (2.2603)

12. Primary Outcome: RSV Viral Load at Day 5
Description: RSV viral load was measured as log10 copies/mL by qRT-PCR assay in the mid-turbinate nasal swab specimens.
Time Frame: Day 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 20 | 21 | 20
Log10 copies/mL | 2.384 (2.4214) | 3.528 (1.9824) | 2.351 (2.1302)

13. Primary Outcome: RSV Viral Load at Day 8
Description: RSV viral load was measured as log10 copies/mL by qRT-PCR assay in the mid-turbinate nasal swab specimens.
Time Frame: Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 18 | 20 | 21
Log10 copies/mL | 0.661 (1.5572) | 1.804 (1.7888) | 1.398 (1.5958)

14. Primary Outcome: RSV Viral Load at Day 14
Description: RSV viral load was measured as log10 copies/mL by qRT-PCR assay in the mid-turbinate nasal swab specimens.
Time Frame: Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 19 | 18 | 19
Log10 copies/mL | 0.421 (1.2601) | 0.290 (0.8579) | 0.492 (0.9910)

15. Primary Outcome: RSV Viral Load at Day 21
Description: RSV viral load was measured as log10 copies/mL by qRT-PCR assay in the mid-turbinate nasal swab specimens.
Time Frame: Day 21
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 20 | 19 | 20
Log10 copies/mL | 0.108 (0.4808) | 0.113 (0.4932) | 0.253 (0.7866)

16. Primary Outcome: Time to Undetectable RSV Viral Load
Description: The time to undetectable nasal RSV RNA viral load was defined as the time in days from initiation of study treatment until first post-baseline time point at which RSV RNA was undetectable and after which time there were no more detectable virus assessments.
Time Frame: Up to Day 21
Population: The ITT-i population consisted of all randomized participants who received at least 1 dose of study drug and who had a central lab-confirmed RSV infection.
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 23 | 21 | 22
Days | 7.0 (5.92) [5.92 to 9.90] | 8.0 (6.86) [6.86 to 12.80] | 9.7 (7.03) [7.03 to 11.74]

17. Primary Outcome: Percentage of Participants With Undetectable RSV Viral Load at Day 3
Description: Percentage of participants with undetectable RSV viral load at Day 3 were reported.
Time Frame: Day 3
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 21 | 20 | 20
Percentage of participants | 28.6 | 5.0 | 20.0

18. Primary Outcome: Percentage of Participants With Undetectable RSV Viral Load at Day 5
Description: Percentage of participants with undetectable RSV viral load at Day 5 were reported.
Time Frame: Day 5
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 20 | 21 | 20
Percentage of participants | 40.0 | 14.3 | 35.0

19. Primary Outcome: Percentage of Participants With Undetectable RSV Viral Load at Day 8
Description: Percentage of participants with undetectable RSV viral load at Day 8 were reported.
Time Frame: Day 8
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 18 | 20 | 21
Percentage of participants | 83.3 | 45.0 | 52.4

20. Primary Outcome: Percentage of Participants With Undetectable RSV Viral Load at Day 14
Description: Percentage of participants with undetectable RSV viral load at Day 14 were reported.
Time Frame: Day 14
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 19 | 18 | 19
Percentage of participants | 89.5 | 88.9 | 78.9

21. Primary Outcome: Percentage of Participants With Undetectable RSV Viral Load at Day 21
Description: Percentage of participants with undetectable RSV viral load at Day 21 were reported.
Time Frame: Day 21
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 19 | 18 | 20
Percentage of participants | 95.0 | 94.7 | 90.0

22. Secondary Outcome: Number of Participants With Adverse Events (AEs) as a Measure of Safety and Tolerability
Description: An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Time Frame: Up to Day 28
Population: The safety analysis set included all participants who received at least 1 dose of study agent, analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 24 | 24 | 24
Participants | 9 | 18 | 15

23. Secondary Outcome: Number of Participants With Worst Treatment-Emergent Laboratory Abnormalities
Description: Number of participants with worst treatment-emergent laboratory abnormalities (serum chemistry, hematology and urinalyses) were reported based on DMID toxicity grading scale. DMID toxicity grade categorized as Grade 1=mild(mild discomfort (< 48 hours); no medical intervention/therapy required), Grade 2= moderate (Moderate Mild to moderate limitation in activity - some assistance may be needed; no or minimal medical intervention/therapy required), Grade 3= severe (severe Marked limitation in activity, some assistance usually required; medical intervention/therapy required, hospitalizations possible), and Grade 4=life threatening (extreme limitation in activity, significant assistance required; significant medical intervention/therapy required, hospitalization or hospice care probable).
Time Frame: Up to Day 28
Population: The safety analysis set included all participants who received at least 1 dose of study agent, analyzed as treated. Here 'N' (number of participants analyzed) signifies number of participants who were valuable for this outcome measure. Here, "n (number analysed)" is defined as number of participants analyzed for specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 22 | 24 | 23
Participants
  Serum chemistry: Alkaline Phosphatase (Grade 1) | 1 | 0 | 1
  Serum chemistry: Alanine Aminotransferase (Grade 1): number analyzed (Participants) | 21 | 24 | 23
  Serum chemistry: Alanine Aminotransferase (Grade 1) | 1 | 0 | 2
  Serum chemistry: Alanine Aminotransferase (Grade 2): number analyzed (Participants) | 21 | 24 | 23
  Serum chemistry: Alanine Aminotransferase (Grade 2) | 0 | 2 | 1
  Serum chemistry: Aspartate Aminotransferase (Grade 1): number analyzed (Participants) | 21 | 24 | 23
  Serum chemistry: Aspartate Aminotransferase (Grade 1) | 1 | 1 | 2
  Serum chemistry: Hyperbilirubinemia (Grade 1) | 1 | 0 | 1
  Serum chemistry: Hyperglycemia (Grade 1) | 4 | 2 | 4
  Serum chemistry: Hyperglycemia (Grade 2) | 0 | 3 | 0
  Serum chemistry: Hypoglycemia (Grade 1) | 0 | 1 | 0
  Serum chemistry: Hyperkalemia (Grade 1) | 0 | 1 | 1
  Serum chemistry: Hypomagnesemia (Grade 1) | 0 | 0 | 1
  Serum chemistry: Hypophosphatemia (Grade 1) | 0 | 1 | 1
  Hypernatremia (Grade 1) | 0 | 0 | 2
  Serum chemistry: Hyperuricemia (Grade 1) | 2 | 3 | 1
  Serum chemistry: Hyperuricemia (Grade 2) | 0 | 1 | 0
  Serum chemistry: Renal Function Creatinine (Grade 1) | 0 | 1 | 0
  Hematology: Hemoglobin (Grade 1) | 1 | 0 | 0
  Hematology: Leukocytes High (Grade 1) | 1 | 0 | 0
  Hematology: Leukocytes High (Grade 2) | 1 | 0 | 0
  Hematology: Leukocytes High (Grade 3) | 1 | 0 | 0
  Hematology: Coagulation Prothrombin Time (Grade 1): number analyzed (Participants) | 22 | 23 | 23
  Hematology: Coagulation Prothrombin Time (Grade 1) | 1 | 0 | 0
  Hematology: Coagulation Prothrombin Time (Grade 2): number analyzed (Participants) | 22 | 23 | 23
  Hematology: Coagulation Prothrombin Time (Grade 2) | 0 | 0 | 2
  Urinalysis: Dipstick Protein (Grade 1): number analyzed (Participants) | 21 | 24 | 23
  Urinalysis: Dipstick Protein (Grade 1) | 0 | 0 | 1
  Urinalysis: Urine (Grade 1): number analyzed (Participants) | 9 | 8 | 9
  Urinalysis: Urine (Grade 1) | 0 | 1 | 1
  Urinalysis Urine (Grade 2): number analyzed (Participants) | 9 | 8 | 9
  Urinalysis Urine (Grade 2) | 1 | 1 | 0

24. Secondary Outcome: Number of Participants With Worst Treatment-Emergent Vital Sign Abnormalities
Description: Number of participants with worst treatment emergent vital sign abnormalities (including Systolic blood pressure [SBP] and diastolic blood pressure [DBP]) as abnormally low, mild increased, moderate increased and severe increased were reported. SBP: Abnormally low- Less than or equal to (<=) 50 mmHg, Grade 1 (mild)- 90 mmHg - < 100 mmHg, Grade 2 (moderate)- greater than or equal to (>=)100 mmHg to < 110 mmHg, Grade 3 (severe)- >=110 mmHg; DBP: Abnormally low- <=90 mmHg, Grade 1 (mild)- 140 mmHg - < 160 mmHg, Grade 2 (moderate)- >=160 mmHg to < 180 mmHg, Grade 3 (severe)- >=180 mmHg.
Time Frame: Up to Day 28
Population: The safety analysis set included all participants who received at least 1 dose of study agent, analyzed as treated. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 23 | 24 | 23
Participants
  Abnormally low DBP | 0 | 0 | 2
  Mild increased DBP | 0 | 3 | 0
  Moderate increased DBP | 1 | 0 | 0
  Abnormally low SBP | 0 | 1 | 1
  Mild increased SBP | 1 | 5 | 3
  Moderate increased SBP | 0 | 0 | 1
  Severe increased SBP | 1 | 0 | 0

25. Secondary Outcome: Number of Participants With Worst Treatment-Emergent (TE) Electrocardiograms (ECGs) Abnormalities
Description: The number of participants with worst TE ECG abnormalities were reported. The ECG variables that were analyzed included heart rate, PR interval, QRS interval, QT interval, and corrected QT (QTc) interval. Parameters for abnormal ECG findings were QT interval corrected for heart rate (QTc) according to Bazett's formula (QTcB or Borderline Prolonged QTcB) Interval ([450 milliseconds {ms}, 480 ms], [480 ms, 500 ms], and [more than 500 ms]), QTc according to Fridericia's formula (QTcF or Borderline Prolonged QTcB) Interval ([450 ms, 480 ms], [480 ms, 500 ms], and [more than 500 ms]).
Time Frame: Up to Day 28
Population: The safety analysis set included all participants who received at least 1 dose of study agent, analyzed as treated. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure. Here, 'n' (number analyzed) signifies number of participants who were analyzed for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 22 | 24 | 23
Participants
  Abnormally low heart rate | 0 | 1 | 1
  Abnormally high PR interval: number analyzed (Participants) | 22 | 24 | 21
  Abnormally high PR interval | 1 | 0 | 0
  Abnormally high QRS interval | 1 | 0 | 0
  QTcB Increase between 30 and 60 ms (Bazett): number analyzed (Participants) | 22 | 23 | 22
  QTcB Increase between 30 and 60 ms (Bazett) | 3 | 1 | 0
  QTcF Increase between 30 and 60 ms (Fridericia): number analyzed (Participants) | 22 | 23 | 22
  QTcF Increase between 30 and 60 ms (Fridericia) | 3 | 0 | 1
  Borderline prolonged QTcB | 5 | 2 | 1
  Borderline prolonged QTcF | 0 | 1 | 0

26. Secondary Outcome: Peripheral Capillary Oxygen Saturation (SpO2) Over Time
Description: Peripheral capillary oxygen saturation was measured by the investigator over time.
Time Frame: Baseline, Days 3, 8, 14, and 21
Population: The ITT-i population consisted of all randomized participants who received at least 1 dose of study drug and who had a central lab-confirmed RSV infection. Here, 'n' (number analyzed) signifies number of participants who were analyzed at specified timepoints. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of SpO2 (%)
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 22 | 21 | 21
Percentage of SpO2 (%)
  Baseline | 95.6 (2.72) | 96.0 (2.60) | 95.8 (2.74)
  Day 3: number analyzed (Participants) | 21 | 21 | 20
  Day 3 | 95.8 (2.62) | 96.8 (2.17) | 95.7 (3.57)
  Day 8: number analyzed (Participants) | 19 | 21 | 21
  Day 8 | 97.2 (1.69) | 96.5 (2.23) | 96.9 (2.26)
  Day 14: number analyzed (Participants) | 20 | 19 | 20
  Day 14 | 97.4 (0.99) | 96.6 (2.14) | 96.7 (1.81)
  Day 21: number analyzed (Participants) | 20 | 19 | 20
  Day 21 | 97.1 (1.23) | 97.1 (1.47) | 96.6 (2.41)

27. Secondary Outcome: Change From Baseline in Peripheral Capillary Oxygen Saturation
Description: Change from baseline in peripheral capillary oxygen saturation levels was calculated by the investigator.
Time Frame: Baseline to Days 3, 8, 14 and 21
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: % of SpO2
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 20 | 21 | 20
% of SpO2
  Baseline to Day 3: number analyzed (Participants) | 20 | 21 | 19
  Baseline to Day 3 | 0.5 (2.21) | 0.9 (1.73) | 0.2 (2.44)
  Baseline to Day 8: number analyzed (Participants) | 18 | 21 | 20
  Baseline to Day 8 | 1.3 (2.72) | 0.5 (1.29) | 1.1 (2.07)
  Baseline to Day 14: number analyzed (Participants) | 19 | 19 | 19
  Baseline to Day 14 | 1.2 (2.10) | 0.7 (1.73) | 1.2 (2.09)
  Baseline to Day 21: number analyzed (Participants) | 19 | 19 | 19
  Baseline to Day 21 | 1.3 (3.11) | 1.2 (2.22) | 1.1 (2.21)

28. Secondary Outcome: Pulse Rate Over Time
Description: Pulse rate was measured by the investigator over time.
Time Frame: Baseline, Days 3, 8, 14 and 21
Population: The ITT-i population consisted of all randomized participants who received at least 1 dose of study drug and who had a central lab-confirmed RSV infection. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure. Here, 'n' (number analyzed) signifies number of participants who were analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: Beats/min
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 23 | 21 | 22
Beats/min
  Baseline | 76.9 (10.86) | 78.0 (12.16) | 77.8 (13.05)
  Day 3: number analyzed (Participants) | 21 | 21 | 20
  Day 3 | 76.4 (11.88) | 76.6 (13.20) | 78.7 (15.64)
  Day 8: number analyzed (Participants) | 19 | 21 | 21
  Day 8 | 70.7 (8.22) | 74.5 (12.74) | 71.8 (10.58)
  Day 14: number analyzed (Participants) | 20 | 19 | 20
  Day 14 | 73.0 (12.62) | 71.4 (13.09) | 73.3 (6.27)
  Day 21: number analyzed (Participants) | 20 | 19 | 20
  Day 21 | 69.4 (7.13) | 71.9 (9.76) | 71.7 (10.00)

29. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Change from baseline in pulse rate was calculated and reported by the investigator.
Time Frame: Baseline to Days 3, 8, 14 and 21
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Beats/min
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 21 | 21 | 21
Beats/min
  Baseline to Day 3: number analyzed (Participants) | 21 | 21 | 20
  Baseline to Day 3 | 0.0 (10.27) | -1.4 (10.17) | 0.2 (11.80)
  Baseline to Day 8: number analyzed (Participants) | 19 | 21 | 21
  Baseline to Day 8 | -5.4 (13.17) | -3.5 (14.03) | -6.4 (11.61)
  Baseline to Day 14: number analyzed (Participants) | 20 | 19 | 20
  Baseline to Day 14 | -4.3 (13.16) | -7.4 (13.76) | -5.3 (10.29)
  Baseline to Day 21: number analyzed (Participants) | 20 | 19 | 20
  Baseline to Day 21 | -6.9 (9.11) | -6.8 (12.11) | -6.9 (12.85)

30. Secondary Outcome: Respiratory Rate Over Time
Description: Respiratory rate was measured by the investigator over time.
Time Frame: Baseline, Days 3, 8, 14 and 21
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Breaths/min
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 23 | 21 | 21
Breaths/min
  Baseline | 18.2 (3.55) | 18.0 (3.08) | 19.2 (3.52)
  Day 3: number analyzed (Participants) | 21 | 21 | 19
  Day 3 | 17.1 (2.64) | 16.7 (3.02) | 18.3 (3.06)
  Day 8: number analyzed (Participants) | 19 | 21 | 21
  Day 8 | 16.9 (1.82) | 17.4 (4.15) | 18.0 (2.48)
  Day 14: number analyzed (Participants) | 20 | 19 | 20
  Day 14 | 16.6 (2.11) | 16.4 (3.10) | 18.1 (2.44)
  Day 21: number analyzed (Participants) | 20 | 19 | 20
  Day 21 | 16.6 (2.23) | 15.7 (3.41) | 17.6 (2.82)

31. Secondary Outcome: Change From Baseline in Respiratory Rate
Description: Change from baseline in respiratory rate was calculated and reported by the investigator.
Time Frame: Baseline to Days 3, 8, 14 and 21
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Breaths/min
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 21 | 21 | 21
Breaths/min
  Baseline to Day 3: number analyzed (Participants) | 21 | 21 | 19
  Baseline to Day 3 | -0.9 (2.10) | -1.3 (3.52) | -0.8 (2.25)
  Baseline to Day 8: number analyzed (Participants) | 19 | 21 | 21
  Baseline to Day 8 | -1.4 (2.34) | -0.6 (4.17) | -1.1 (3.51)
  Baseline to Day 14: number analyzed (Participants) | 20 | 19 | 20
  Baseline to Day 14 | -1.8 (2.83) | -1.7 (3.59) | -1.3 (3.33)
  Baseline to Day 21: number analyzed (Participants) | 20 | 19 | 20
  Baseline to Day 21 | -1.8 (2.73) | -2.4 (4.34) | -1.8 (3.33)

32. Secondary Outcome: Body Temperature Over Time
Description: Body temperature was measured over time. Participants were provided a thermometer and asked to record body temperature in the electronic device.
Time Frame: Baseline, Days 3, 8, 14 and 21
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 23 | 21 | 22
degree Celsius
  Baseline | 36.83 (0.622) | 36.73 (0.601) | 36.75 (0.561)
  Day 3: number analyzed (Participants) | 21 | 20 | 21
  Day 3 | 36.57 (0.572) | 36.65 (0.574) | 36.69 (0.446)
  Day 8: number analyzed (Participants) | 18 | 21 | 20
  Day 8 | 36.26 (0.396) | 36.44 (0.527) | 36.55 (0.404)
  Day 14: number analyzed (Participants) | 20 | 19 | 20
  Day 14 | 36.37 (0.389) | 36.38 (0.346) | 36.50 (0.291)
  Day 21: number analyzed (Participants) | 20 | 19 | 20
  Day 21 | 36.32 (0.380) | 36.40 (0.380) | 36.46 (0.299)

33. Secondary Outcome: Change From Baseline in Body Temperature
Description: Change from baseline in body temperature was calculated and reported. Participants were provided a thermometer and asked to record body temperature in the electronic device.
Time Frame: Baseline to Days 3, 5, 8, 14 and 21
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 21 | 21 | 21
degree Celsius
  Baseline to Day 3: number analyzed (Participants) | 21 | 20 | 21
  Baseline to Day 3 | -0.27 (0.390) | -0.11 (0.621) | -0.01 (0.595)
  Baseline to Day 5: number analyzed (Participants) | 19 | 21 | 19
  Baseline to Day 5 | -0.63 (0.667) | -0.41 (0.645) | -0.17 (0.650)
  Baseline to Day 8: number analyzed (Participants) | 18 | 21 | 20
  Baseline to Day 8 | -0.55 (0.465) | -0.29 (0.652) | -0.11 (0.477)
  Baseline to Day 14: number analyzed (Participants) | 20 | 19 | 20
  Baseline to Day 14 | -0.48 (0.402) | -0.40 (0.624) | -0.20 (0.411)
  Baseline to Day 21: number analyzed (Participants) | 20 | 19 | 20
  Baseline to Day 21 | -0.52 (0.537) | -0.37 (0.615) | -0.24 (0.503)

34. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Point 0 Hours Until 24 Hours Post Dose
Description: AUC (0-24) is defined as area under the plasma concentration-time curve from time point 0 hours until 24 hours post dose.
Time Frame: 0 to 24 hours post dose on Days 1 and 7
Population: Pharmacokinetic (PK) analysis set included all participants who received JNJ-53718678 and for whom at least one PK concentration was reported. Here, 'n' (number analyzed) signifies number of participants who were analyzed at specified timepoints. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanograms*hours per milliliter (ng*h/mL)
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo
Number analyzed (Participants) | 16 | 18
nanograms*hours per milliliter (ng*h/mL)
  Day 1: number analyzed (Participants) | 15 | 17
  Day 1 | 29800 (9180) | 4530 (1560)
  Day 7 | 41200 (15300) | 5470 (1620)

35. Secondary Outcome: Severity of Signs and Symptoms of RSV Assessed by Respiratory Infection-Patient Reported Outcomes (RI-PRO) Questionnaire
Description: The severity of signs and symptoms of RSV infection was assessed using the RI-PRO questionnaire. The RI-PRO questionnaire is 32-item questionnaire. It summarizes severity of 6 symptom domains: nose (4 items), throat (3 items), eyes (3 items), chest/respiratory (7 items), gastrointestinal (4 items), and body/systemic (11 items). Each RI-PRO domain score ranges from 0 (symptom free) to 4 (very severe symptoms). Domain scores were calculated as the arithmetic mean of the scores for items within the domain.
Time Frame: Baseline, Days 3, 5, 8, 14 and 21
Population: The ITT-i population consisted of all randomized participants who received at least 1 dose of study drug and who had a central lab-confirmed RSV infection. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure. Here, 'n' (number analyzed) signifies number of participants who were analyzed at specified timepoints for specified categories.
Measure: Mean (Standard Deviation); unit: Scale on a score
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 21 | 21 | 22
Scale on a score
  Nose: Baseline | 2.32 (0.912) | 2.16 (0.816) | 1.91 (0.9990)
  Nose: Day 3: number analyzed (Participants) | 19 | 18 | 19
  Nose: Day 3 | 1.84 (0.983) | 1.01 (0.720) | 1.25 (0.182)
  Nose: Day 5: number analyzed (Participants) | 18 | 19 | 16
  Nose: Day 5 | 1.11 (0.614) | 0.63 (0.591) | 0.94 (0.649)
  Nose: Day 8: number analyzed (Participants) | 20 | 21 | 17
  Nose: Day 8 | 0.88 (0.676) | 0.45 (0.557) | 0.68 (0.630)
  Nose: Day 14: number analyzed (Participants) | 18 | 19 | 17
  Nose: Day 14 | 0.43 (0.561) | 0.20 (0.504) | 0.38 (0.580)
  Nose: Day 21: number analyzed (Participants) | 14 | 14 | 12
  Nose: Day 21 | 0.45 (0.674) | 0.18 (0.532) | 0.48 (0.607)
  Throat: Baseline: number analyzed (Participants) | 21 | 20 | 22
  Throat: Baseline | 1.46 (1.142) | 2.02 (1.197) | 1.36 (1.186)
  Throat: Day 3: number analyzed (Participants) | 19 | 18 | 19
  Throat: Day 3 | 1.02 (0.828) | 0.78 (0.741) | 0.67 (0.720)
  Throat: Day 5: number analyzed (Participants) | 18 | 19 | 16
  Throat: Day 5 | 0.74 (0.813) | 0.44 (0.485) | 0.33 (0.471)
  Throat: Day 8: number analyzed (Participants) | 20 | 21 | 17
  Throat: Day 8 | 0.13 (0.274) | 0.22 (0.355) | 0.25 (0.417)
  Throat: Day 14: number analyzed (Participants) | 18 | 19 | 17
  Throat: Day 14 | 0.00 (0.000) | 0.02 (0.076) | 0.18 (0.393)
  Throat: Day 21: number analyzed (Participants) | 14 | 14 | 12
  Throat: Day 21 | 0.02 (0.089) | 0.00 (0.00) | 0.19 (0.388)
  Eye: Baseline: number analyzed (Participants) | 21 | 20 | 22
  Eye: Baseline | 0.97 (1.115) | 0.80 (0.847) | 1.17 (0.821)
  Eye: Day 3: number analyzed (Participants) | 19 | 18 | 19
  Eye: Day 3 | 0.77 (0.802) | 0.26 (0.421) | 0.65 (0.662)
  Eye: Day 5: number analyzed (Participants) | 18 | 19 | 16
  Eye: Day 5 | 0.46 (0.742) | 0.14 (0.339) | 0.50 (0.798)
  Eye: Day 8: number analyzed (Participants) | 20 | 21 | 17
  Eye: Day 8 | 0.13 (0.251) | 0.08 (0.296) | 0.35 (0.629)
  Eye: Day 14: number analyzed (Participants) | 18 | 19 | 17
  Eye: Day 14 | 0.07 (0.244) | 0.04 (0.153) | 0.29 (0.406)
  Eye: Day 21: number analyzed (Participants) | 14 | 14 | 12
  Eye: Day 21 | 0.00 (0.00) | 0.00 (0.00) | 0.39 (0.529)
  Chest/Respiratory: Baseline: number analyzed (Participants) | 21 | 20 | 22
  Chest/Respiratory: Baseline | 1.86 (0.804) | 1.96 (0.815) | 1.74 (0.659)
  Chest/Respiratory: Day 3: number analyzed (Participants) | 19 | 18 | 19
  Chest/Respiratory: Day 3 | 1.46 (0.704) | 1.37 (0.750) | 1.37 (0.715)
  Chest/Respiratory: Day 5: number analyzed (Participants) | 18 | 19 | 16
  Chest/Respiratory: Day 5 | 1.02 (0.542) | 0.95 (0.767) | 1.12 (0.648)
  Chest/Respiratory: Day 8: number analyzed (Participants) | 20 | 21 | 17
  Chest/Respiratory: Day 8 | 0.69 (0.579) | 0.72 (0.632) | 0.81 (0.616)
  Chest/Respiratory: Day 14: number analyzed (Participants) | 18 | 19 | 17
  Chest/Respiratory: Day 14 | 0.40 (0.494) | 0.31 (0.566) | 0.53 (0.599)
  Chest/Respiratory: Day 21: number analyzed (Participants) | 14 | 14 | 12
  Chest/Respiratory: Day 21 | 0.28 (0.607) | 0.32 (0.666) | 0.60 (0.523)
  Gastrointestinal: Baseline: number analyzed (Participants) | 21 | 20 | 22
  Gastrointestinal: Baseline | 0.17 (0.398) | 0.38 (0.666) | 0.26 (0.426)
  Gastrointestinal: Day 3: number analyzed (Participants) | 19 | 18 | 19
  Gastrointestinal: Day 3 | 0.72 (0.986) | 0.47 (0.712) | 0.50 (0.692)
  Gastrointestinal: Day 5: number analyzed (Participants) | 18 | 19 | 16
  Gastrointestinal: Day 5 | 0.40 (0.648) | 0.36 (0.385) | 0.48 (0.559)
  Gastrointestinal: Day 8: number analyzed (Participants) | 20 | 21 | 17
  Gastrointestinal: Day 8 | 0.24 (0.425) | 0.19 (0.249) | 0.28 (0.423)
  Gastrointestinal: Day 14: number analyzed (Participants) | 18 | 19 | 17
  Gastrointestinal: Day 14 | 0.08 (0.354) | 0.01 (0.057) | 0.07 (0.212)
  Gastrointestinal: Day 21: number analyzed (Participants) | 14 | 14 | 12
  Gastrointestinal: Day 21 | 0.02 (0.067) | 0.00 (0.00) | 0.17 (0.268)
  Body/Systemic: Baseline: number analyzed (Participants) | 21 | 20 | 22
  Body/Systemic: Baseline | 1.47 (0.925) | 1.50 (0.649) | 1.34 (0.770)
  Body/Systemic: Day 3: number analyzed (Participants) | 19 | 18 | 19
  Body/Systemic: Day 3 | 1.02 (0.748) | 0.55 (0.435) | 0.82 (0.633)
  Body/Systemic: Day 5: number analyzed (Participants) | 18 | 19 | 16
  Body/Systemic: Day 5 | 0.54 (0.429) | 0.37 (0.442) | 0.61 (0.463)
  Body/Systemic: Day 8: number analyzed (Participants) | 20 | 21 | 17
  Body/Systemic: Day 8 | 0.20 (0.368) | 0.27 (0.296) | 0.36 (0.471)
  Body/Systemic: Day 14: number analyzed (Participants) | 18 | 19 | 17
  Body/Systemic: Day 14 | 0.18 (0.281) | 0.10 (0.186) | 0.36 (0.480)
  Body/Systemic: Day 21: number analyzed (Participants) | 14 | 14 | 12
  Body/Systemic: Day 21 | 0.17 (0.300) | 0.09 (0.147) | 0.27 (0.384)

36. Secondary Outcome: Duration of Signs and Symptoms of RSV Assessed by RI-PRO
Description: Duration of signs and symptoms of RSV infection was assessed by the time to resolution of all RSV symptoms from RI-PRO questionnaire. Resolution was defined as a score of 'Not at all/symptom-free' (score=0) or 'A little bit' (score=1) for at least 24 hours. The RI-PRO questionnaire is a 32-item questionnaire. It summarizes severity of 6 symptom domains: nose (4 items), throat (3 items), eyes (3 items), chest/respiratory (7 items), gastrointestinal (4 items) and body/systemic (11 items). Each RI-PRO score ranges from 0 (symptom-free) to 4 (very severe symptoms).
Time Frame: Baseline up to Day 21
Population: as for outcome 2
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 20 | 20 | 20
days | 7.9 [6.90 to 18.92] | 7.4 [5.05 to 9.52] | 15.9 [6.40 to NA] — Here, NA signifies that upper bound of the 90% confidence interval could not be calculated due to the low number of participants and censoring.

37. Secondary Outcome: Time to Resolution of Key RSV Symptoms as Assessed by RI-PRO Questionnaire
Description: Time to resolution of key RSV symptoms (congested or stuffy nose, sore or painful throat, trouble breathing, chest tightness, coughing, coughed up mucus or phlegm, weak or tired) as assessed by RI-PRO questionnaire was reported. Resolution of RSV symptoms was defined as a score of 'Not at all/symptom free' (score = 0) or 'A little bit' (score = 1) for at least 24 hours for symptoms of the RI-PRO questionnaire. The RI-PRO questionnaire is 32-item questionnaire. It summarizes severity of 6 symptom domains: nose (4 items), throat (3 items), eyes (3 items), chest/respiratory (7 items), gastrointestinal (4 items), and body/systemic (11 items). Each RI-PRO score ranges from 0 (symptom-free) to 4 (very severe symptoms).
Time Frame: Up to Day 21
Population: as for outcome 2
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 22 | 21 | 22
Days | 7.1 [5.03 to 11.43] | 7.6 [5.93 to 8.32] | 9.6 [5.95 to 14.0]

38. Secondary Outcome: Time to Return to Usual Activity/Health Based on RI-PRO Questionnaire
Description: Time from the first dose of study drug until the time to return to usual activity/health was determined. Return to usual activity/health when the response is 'Yes' on RI-PRO additional question 7 ('Have you returned to your usual activity/health today?') for at least 24 hours.
Time Frame: Up to Day 21
Population: as for outcome 16
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
Number analyzed (Participants) | 23 | 21 | 22
days
  Time to return to usual activity | 6.0 (2.99) [2.99 to 8.33] | 3.0 (1.39) [1.39 to 7.88] | 5.6 (4.62) [4.62 to 10.62]
  Time to return to usual health | 8.3 (5.51) [5.51 to 11.87] | 8.6 (5.57) [5.57 to 10.81] | 9.1 (5.62) [5.62 to 10.64]

39. Secondary Outcome: Predose Plasma Concentration (Ctrough) of JNJ-53718678
Description: Ctrough is the trough plasma concentration of JNJ-53718678 estimated by population PK model.
Time Frame: Predose on Days 1 and 7
Population: PK analysis set included all participants who received JNJ-53718678 and for whom at least one PK concentration was reported. Here, 'n' (number analyzed) signifies number of participants who were analyzed at specified timepoints. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo
Number analyzed (Participants) | 16 | 18
nanograms per milliliter (ng/mL)
  Day 1: number analyzed (Participants) | 15 | 17
  Day 1 | 514 (249) | 68.2 (36.2)
  Day 7 | 774 (451) | 84.4 (39.4)

40. Secondary Outcome: Maximum Plasma Concentration (Cmax) of JNJ-53718678
Description: Cmax is the maximum plasma concentration of JNJ-53718678 estimated by population PK model.
Time Frame: Days 1 and 7
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo
Number analyzed (Participants) | 17 | 20
ng/mL
  Day 1 | 2870 (802) | 490 (150)
  Day 7: number analyzed (Participants) | 16 | 18
  Day 7 | 3540 (1050) | 552 (131)

ADVERSE EVENTS:
Time Frame: Up to Day 28
Description: The safety analysis set included all participants who received at least 1 dose of study agent, analyzed as treated.
Arm/Group | Treatment A: JNJ-53718678 500 mg | Treatment B: JNJ-53718678 80 mg + Placebo | Treatment C: Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 6/24 | 13/24 | 11/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A: JNJ-53718678 500 mg (N=24) | Treatment B: JNJ-53718678 80 mg + Placebo (N=24) | Treatment C: Placebo (N=24)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 9 (14) | 9 (10)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
The Respiratory Infection Intensity and Impact Questionnaire (RiiQ) Scale that replaced Respiratory Infection-Patient Reported Outcomes (RI-PRO) questionnaire was only evaluated in the 5 participants who were enrolled after implementation of protocol amendment 1. This sample size was too small to draw conclusions on comparison between RiiQ and RI-PRO results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will with hold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/75/NCT03379675/Prot_002.pdf
  • Statistical Analysis Plan (2019-09-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT03379675/SAP_003.pdf